CLINICAL TRIAL: NCT07105475
Title: Randomized, Sham Controlled Study for the Treatment of ADHD Using High and Low Frequency Paired Associative Deep Transcranial Magnetic Stimulation
Brief Title: Treatment of ADHD Using High and Low Frequency Paired Associative Deep Transcranial Magnetic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Zachary Katz, Principal Investigator, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0152-23-SOR
Record Dates: First submitted 2025-07-13; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Neurodevelopmental Disorders; Prefrontal Cortex Dysregulation; Cortical Arousal Imbalance
Keywords: ADHD; Transcranial Magnetic Stimulation (TMS); Paired Associative Stimulation (PAS); Prefrontal Cortex; Hemispheric Asymmetry
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Low-Frequency Active PAS Treatment (ADHD Patients) (Experimental): Participants in this group will undergo three weeks of low-frequency paired associative stimulation (PAS) treatment. This involves the application of TMS at a low frequency to stimulate brain areas, specifically targeting the prefrontal cortex, to potentially improve symptoms of ADHD. The treatment will be administered five days a week for three weeks.
  Interventions: Device: Paired Associative Transcranial Magnetic Stimulation (TMS)
- High-Frequency Active PAS Treatment (ADHD Patients) (Experimental): Participants in this group will receive three weeks of high-frequency PAS treatment. High-frequency TMS will be applied to stimulate brain areas, particularly the prefrontal cortex, to enhance cortical arousal and improve ADHD symptoms. This treatment will also be administered five days a week for three weeks.
  Interventions: Device: Paired Associative Transcranial Magnetic Stimulation (TMS)
- Low-Frequency Sham PAS Treatment (ADHD Patients) (Placebo Comparator): This group will undergo three weeks of sham PAS treatment, where the procedure mimics the active treatment but with the magnetic stimulation at a minimal power (20% of the subject's motor threshold). The goal is to serve as a placebo control to evaluate the effectiveness of the active treatments. This sham treatment will be administered five days a week for three weeks.
  Interventions: Device: Paired Associative Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Paired Associative Transcranial Magnetic Stimulation (TMS) — Transcranial Magnetic Stimulation (TMS) is a non-invasive technique that uses magnetic fields to stimulate nerve cells in the brain. By placing a coil on the scalp, TMS generates magnetic pulses that induce electrical currents in specific brain regions. This can alter brain activity and potentially influence behavior and symptoms of various neurological and psychiatric conditions.
  PAS involves the use of transcranial magnetic stimulation (TMS) at a low and high frequency to stimulate the prefrontal cortex at different areas of the brain. The goal is to assess its effects on cortical arousal and ADHD symptoms. Participants will receive daily sessions of this stimulation for three weeks, with the stimulation designed to influence brain activity and potentially alleviate symptoms of ADHD.
  Other Names: Low-Frequency Paired Associative Stimulation (PAS); High-Frequency Paired Associative Stimulation (PAS)

SUMMARY:
This study investigates the effects of high and low-frequency paired associative deep transcranial magnetic stimulation (dTMS) on adults with Attention Deficit Hyperactivity Disorder (ADHD). The study aims to explore whether targeting the prefrontal cortex with paired stimulation can improve symptoms of ADHD by balancing cortical arousal between the brain hemispheres. A total of 90 participants with ADHD will be recruited. Participants with ADHD will undergo three weeks of daily TMS treatment, while participants who receive a sham treatment will be included for baseline comparisons. The study will measure electrophysiological, cognitive, and clinical outcomes using a variety of assessments, including EEG, cognitive tests, and CAARS to evaluate the treatment's efficacy.

DETAILED DESCRIPTION:
Introduction Transcranial Magnetic Stimulation (TMS) is a non-invasive technique that uses magnetic fields to stimulate nerve cells in the brain, potentially altering brain activities and influencing behavior. It has been applied in both healthy individuals and patients to study brain activity, behavior, and therapeutic effects. TMS can be administered as single pulses or repetitive stimuli, with the latter showing lasting effects beyond the treatment session. High-frequency TMS is FDA-approved for treating major depressive disorder, obsessive-compulsive disorder, and smoking cessation.

ADHD is a neurodevelopmental disorder characterized by inattention, impulsivity, and hyperactivity. Neuroimaging studies have identified deficits in brain regions such as the prefrontal cortex, basal ganglia, and cerebellum in ADHD patients. Enhancing activity in these areas, particularly the prefrontal cortex, through high-frequency TMS has shown promise in reducing ADHD symptoms.

Research Question and Hypothesis The study aims to assess the effectiveness of paired associative stimulation (PAS) in treating ADHD. It hypothesizes that right-to-left prefrontal paired stimulation can enhance cortical arousal and provide symptom relief. The study includes two active treatment groups (high and low-frequency PAS) and a sham treatment group, with secondary goals to quantify short- and long-term changes in behavior, brain function, and structure.

Methods

Participants Total: 90 ADHD patients ADHD patients: Pre-screened by a psychiatrist; will undergo three weeks of treatment.

Healthy controls: Single session to measure brain activity and arousal.

Length of Experiment Recruitment duration: Approximately three years to recruit 90 ADHD subjects. Individual participation: Three weeks of treatment, with follow-up sessions at one and two months post-treatment.

Procedure Patient recruitment: Includes medical screening, consent, physical and neurological examinations, and psychological assessments.

Experimental Groups:

Group A: Low-frequency active PAS (30 ADHD subjects). Group B: High-frequency active PAS (30 ADHD subjects). Group C: Low-frequency sham PAS (30 ADHD subjects).

Daily Magnetic Therapy Phase 15 TMS treatments over three weeks for ADHD subjects, including cognitive exercises post-TMS. Data collection includes EEG recordings, cognitive tests, and brain response measurements before and after TMS.

Follow-up Phase Two sessions, four weeks apart, assessing treatment effectiveness and side effects through EEG and questionnaires.

Conclusion This study explores the potential of high and low-frequency paired associative dTMS in treating ADHD by targeting interhemispheric balance in the prefrontal cortex. The research will provide insights into the efficacy of PAS as an innovative treatment approach for ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 21-65.
* Aligned with the diagnosis of ADHD according to the criteria of the DSM-5.
* Participants taking medication for the treatment of attention deficit hyperactivity disorder will be asked, starting one week before the start of the treatment until the end, to take Ritalin IR 10mg (provided that the taking of the medication will be done at least 8 hours before the start of the treatment or at least one hour after it. This instruction is also valid for taking the medication on the days of the follow-up sessions (4 and 8 weeks from the end of the daily treatment phase). Ritalin is given as the only option because a drug with a short half-life is needed. The dose can be increased up to 20 mg per dose). The choice of this drug is to ensure that changes in brain function/activity are not the result of the Ritalin medication but of the research intervention.
* Give their written and oral consent to participate in the study.

Exclusion Criteria:

* Additional active psychiatric disorders in Axis I of the DSM-5.
* Antipsychotic treatment, antidepressants, or mood stabilizers.
* History of intolerance to TMS.
* Diagnosis of severe personality disorder according to the DSM-5.
* Current suicidal tendency.
* High and uncontrolled blood pressure.
* History of epilepsy, seizures or febrile seizures.
* History of epilepsy or seizures in first degree relatives.
* History of a head injury or major stroke that produced impairment.
* History of metal in the head (outside the oral cavity).
* History of surgery involving metal implants or a known history of metal particles in the eye, pacemakers, hearing aid implantation, use of neurostimulators, or any medical pump.
* History of drug or alcohol addiction.
* Inability to adequately communicate with the examiner.
* Participation in another medical study at the time of conducting the experiment or 3 months before it.
* Inability of the subject to sign a consent form.
* Pregnancy or not giving a commitment not to get pregnant during the study period or having sex without using contraceptives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD Symptoms Assessed by the Conners' Adult ADHD Rating Scale (CAARS) | Pre-treatment (baseline) and post-treatment assessments at the end of the 3-week treatment phase, with follow-up assessments at 1 month and 2 months after treatment to evaluate sustained symptom improvement.
  This measure evaluates the change in ADHD symptom severity using the Conners' Adult ADHD Rating Scale (CAARS), a standardized and validated assessment tool. The CAARS provides subscale scores (e.g., Inattention, Hyperactivity-Impulsivity, ADHD Index) on a scale ranging from 0 to 100, with higher scores indicating greater symptom severity. Change will be assessed by comparing scores obtained at baseline (pre-treatment) and following the intervention (post-treatment), as well as at 1-month and 2-month follow-up visits.
Change in Cognitive Control Assessed by Stroop Task Performance | Pre-treatment (baseline) and post-treatment (immediately after the 3-week treatment phase). Additional assessments may be conducted during follow-up sessions at 1 month and 2 months after treatment.
  This measure assesses changes in participants' cognitive control by comparing pre-treatment and post-treatment performance on the Stroop Task. Performance is evaluated based on reaction time (milliseconds) and accuracy (% correct responses) in congruent and incongruent trials. Lower reaction times and higher accuracy typically indicate better cognitive control, but outcome-neutral interpretation will be used to assess change.
Change in Working Memory Assessed by N-back Task Performance | Pre-treatment (baseline) and post-treatment (immediately after the 3-week treatment phase). Additional assessments may be conducted during follow-up sessions at 1 month and 2 months after treatment.
  This measure evaluates working memory by comparing participants' pre-treatment and post-treatment performance on the N-back task (2-back condition). Performance is quantified by reaction time (milliseconds) and accuracy (% correct target detections). Lower reaction times and higher accuracy reflect stronger working memory performance, but results will be analyzed in a directionally neutral manner.
Change in EEG Power Spectral Density Across Frequency Bands | Baseline (pre/post Session 1), end of treatment (pre/post Session 15), and at 1-month and 2-month follow-ups. EEG is recorded during rest, cognitive tasks, TMS, TEP, and post-treatment rest at each time point.
  This outcome assesses changes in EEG power spectral density (PSD) in the delta (0.5-4 Hz), theta (4-7 Hz), alpha (8-12 Hz), and beta (13-30 Hz) frequency bands during resting-state EEG. PSD will be calculated using Fourier-based spectral analysis and reported in microvolts squared per hertz (µV²/Hz) at frontal and motor cortex sites.
Change in Raw EEG Voltage | Baseline (pre/post Session 1), end of treatment (pre/post Session 15), and at 1-month and 2-month follow-ups. EEG is recorded during rest, cognitive tasks, TMS, TEP, and post-treatment rest at each time point.
  This outcome measures the overall amplitude of raw EEG signals recorded at rest. Changes in baseline EEG voltage levels will be evaluated across treatment sessions and follow-ups to assess general cortical excitability. Unit of Measure:
  Microvolts (µV).

SECONDARY OUTCOMES:
Long-Term Change in ADHD Symptoms Assessed at Follow-Up by Conners' Adult ADHD Rating Scale (CAARS) | Assessed during follow-up sessions at 1 month and 2 months after the end of the 3-week treatment phase to evaluate the persistence of treatment effects.
  This outcome assesses the persistence of treatment-related changes in ADHD symptoms using the Conners' Adult ADHD Rating Scale (CAARS). The CAARS includes multiple subscale scores (e.g., Inattention, Hyperactivity-Impulsivity) ranging from 0 to 100, with higher scores indicating greater symptom severity. Scores will be compared between post-treatment and follow-up time points to evaluate sustained changes. Unit of Measure: CAARS Subscale Score (0-100).
Long-Term Change in Cognitive Control Assessed at Follow-Up by Stroop Task Performance | Assessed during follow-up sessions at 1 month and 2 months after the end of the 3-week treatment phase to evaluate the persistence of treatment effects.
  This outcome evaluates long-term effects of TMS on cognitive control using the Stroop Task. Performance will be measured by reaction time (milliseconds) and accuracy (% correct responses) during congruent and incongruent trials. Comparisons will be made between post-treatment and follow-up time points to assess sustained changes in executive function. Unit of Measure: Milliseconds (reaction time), Percent correct (% accuracy).
Long-Term Change in Working Memory Assessed at Follow-Up by N-back Task Performance | Assessed during follow-up sessions at 1 month and 2 months after the end of the 3-week treatment phase to evaluate the persistence of treatment effects.
  This outcome evaluates the persistence of treatment-related changes in working memory using the 2-back condition of the N-back Task. Performance will be assessed based on reaction time (milliseconds) and accuracy (% correct target detections). Results from post-treatment and follow-up assessments will be compared. Unit of Measure: Milliseconds (reaction time), Percent correct (% accuracy).
Change in Amplitude of TMS-Evoked Potential (TEP) Components | Baseline (pre/post Session 1), end of treatment (pre/post Session 15), and at 1-month and 2-month follow-ups. EEG is recorded during rest, cognitive tasks, TMS, TEP, and post-treatment rest at each time point.
  This outcome assesses the amplitude of specific TMS-evoked potential (TEP) components (e.g., P30, N45, N100) extracted from EEG data recorded during TMS stimulation sessions. These components reflect cortical excitability and inhibition. Unit of Measure: Microvolts (µV).
Change in Variance of TMS-Evoked Potentials (TEPs) | Baseline (pre/post Session 1), end of treatment (pre/post Session 15), and at 1-month and 2-month follow-ups. EEG is recorded during rest, cognitive tasks, TMS, TEP, and post-treatment rest at each time point.
  This outcome quantifies the trial-by-trial variability of TEP responses to assess consistency of cortical reactivity. Variance in EEG response to TMS will be calculated for each major TEP component. Unit of Measure: Microvolts squared (µV²).
Change in EEG Frequency Characteristics | Baseline (pre/post Session 1), end of treatment (pre/post Session 15), and at 1-month and 2-month follow-ups. EEG is recorded during rest, cognitive tasks, TMS, TEP, and post-treatment rest at each time point.
  This outcome tracks shifts in peak and dominant frequency within delta, theta, alpha, and beta bands during resting EEG. It provides insight into general neurophysiological state and functional changes over time. Unit of Measure: Hertz (Hz).

OTHER OUTCOMES:
Incidence of Adverse Events Reported During and After TMS Treatment | Monitored throughout the 3-week treatment, with documentation of any adverse effects during each treatment session. Follow-up assessments at 1 month and 2 months post-treatment will monitor for any delayed side effects or long-term tolerability issues.
  Adverse events (AEs) will be monitored and documented throughout the TMS intervention and follow-up periods. AEs will be identified using a structured adverse event reporting form completed by study staff during each session and follow-up. Events will be categorized by severity (mild, moderate, severe) and by relation to the intervention (definitely, possibly, or not related). Each participant's number and type of AEs will be recorded. Unit of Measure: Number of adverse events per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Zangen, Study Director — Ben-Gurion University of the Negev; Hadar Shalev, Principal Investigator — Soroka University Medical Center
Locations (1):
- Ben Gurion University of the Negev, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No